CLINICAL TRIAL: NCT05147857
Title: Dilapan Versus Prostaglandin E1 in Induction of Midtrimester Abortion
Brief Title: Mid Trimester Abortion Effectiveness by Dilapan s
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Reem Nasr Abd el hafez Nasr, Principal investigator, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTD
Record Dates: First submitted 2021-11-10; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Abortion Early
Keywords: Abortion; Dilapan s
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesotac in mid trimester (Active Comparator): Prostaglandin
  Interventions: Drug: Misoprostol
- Dilapan s in mid trimester (Active Comparator): is an osmotic hygroscopic dilator produced from a patented Aquacryl® hydrogel that guarantees consistency of action.
  It is a rigid gel rod that increases in volume by absorbing fluids from the cervical canal, so it gradually dilates the cervix The thin 4 mm rod can expand up to 15 mm over a 12-24 hours period. This allows it to dilate and soften the cervix gradually.
  Interventions: Device: Dilapan s

INTERVENTIONS:
Device: Dilapan s — is an osmotic hygroscopic dilator produced from a patented Aquacryl® hydrogel that guarantees consistency of action.
  It is a rigid gel rod that increases in volume by absorbing fluids from the cervical canal, so it gradually dilates the cervix The thin 4 mm rod can expand up to 15 mm over a 12-24 hours period. This allows it to dilate and soften the cervix gradually.
  Arms: Dilapan s in mid trimester
Drug: Misoprostol — Misoprostol is a synthetic prostaglandin medication used to prevent and treat stomach and duodenal ulcers, induce labor, cause an abortion, and treat postpartum bleeding due to poor contraction of the uterus. Misoprostol is taken by mouth when used to prevent gastric ulcers in persons taking NSAIDs.
  Other Names: Misotac
  Arms: Mesotac in mid trimester

SUMMARY:
This study is done aiming to find out an effective method to induce second trimester abortion within a reasonable time and with the least possible cost and complications.

DETAILED DESCRIPTION:
od complete history taking and examination will be performed including measurement of blood pressure, pulse and temperature. Skin was examined for petichae or ecchymosis to exclude coagulation defects or blood diseases. The abdominal examination included detection of the size of the uterus (in cm above symphysis pubis), presence of scar of previous laparotomy, tenderness or rigidity. The local examination included detection of uterine size by bimanual examination, cervical dilatation, consistency, effacement, and position.

Each patient was investigated for hemoglobin content, Rh-typing, blood sugar level, Coagulation profile, renal function tests, and liver function tests.

Our patients were divided into 2 groups, each containing-- patients: In the First group, induction of abortion was carried out by prostaglandin E1 methyl analogue, Misoprestol. It was given by vaginal routeIn the second group, induction of abortion will be started with Dilapan.s followed by surgical evacuation In the First group, the initial Bishop score will be recorded and the minimal dose of one tablet was inserted deep in the posterior fornix. The dose will be repeated every 4 hours till the products of conception are expelled. If remnants of conception are retained for more than 30 minutes, oxytocin drip will be initiated starting with a minimal dose of 2.5 U in 500-ml glucose 5%. Failure of induction was considered if uterine contractions and start of expulsion had not occurred within 36 hours from initiation of therapy.

In the second group, The vagina will be prepared with Povidine iodine as an antiseptic, which is also used to moisten the dilators. A sterile speculum will be inserted and after inspection of the cervix, the anterior lip will stabilized with ring forceps. Using gentle traction on the cervix, the Dilapan dilator will be inserted into the cervical canal, the upper vagina will then packed with a sterile gauze to maintain the dilator in place. The dilators were left for a period not less than 6 and not more than 24 hours. After removal of the gauze, the Dilapan handle will be grasped with forceps and removed with gentle steady downward traction on Dialpan loop itself. The cervical dilatation will be measured by Hegar's dilators and recorded. Surgical evacuation will then carried out under general anesthesia. In cases with gestational age more than 16 weeks, an oxytocin infusion will be MasterDegreeThesis/MFA/ISRO/FacultyOfMedicine/ASU Page 4

added to induce uterine contractions and expulsion of the contents. Failure was considered if dilatation of the cervix was not achieved, or if there was no response to oxytocin within 36 hours.

Clinical data were recorded in an investigative report form and Sudent's (t) test was used to compare means, P value of < 0.05 was considered significant.

ELIGIBILITY:
Inclusion Inclusion Criteria:

* Sure indication of abortion.
* Estimated gestational age between 12-24 weeks as calculated from last normal menstrual period (LNMP) and confirmed by abdominal ultrasound.
* Intact membranes.
* No medical disorder prevents the usage of any of the medications in the study.

Exclusion Criteria:

* History of cervical surgery or presence of cervical scarring.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Abortion | 24 hour from procedure
  Abortion time in days

SECONDARY OUTCOMES:
Hospital stay | 24 hour from admission
  Number of days of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Salma Nassar, MD, Study Director — Ainshams maternity hospital; Ayman Abo nour, Prof, Principal Investigator — Ainshams maternity hospital
Locations (1):
- Ainshams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones RK, Kooistra K. Abortion incidence and access to services in the United States, 2008. Perspect Sex Reprod Health. 2011 Mar;43(1):41-50. doi: 10.1363/4304111. Epub 2011 Jan 10. PMID 21388504
- [Result] Pazol K, Creanga AA, Zane SB, Burley KD, Jamieson DJ; Centers for Disease Control and Prevention (CDC). Abortion surveillance--United States, 2009. MMWR Surveill Summ. 2012 Nov 23;61(8):1-44. PMID 23169413
- [Result] Johnson MR, Riddle AF, Grudzinskas JG, Sharma V, Collins WP, Nicolaides KH. Reduced circulating placental protein concentrations during the first trimester are associated with preterm labour and low birth weight. Hum Reprod. 1993 Nov;8(11):1942-7. doi: 10.1093/oxfordjournals.humrep.a137965. PMID 7507132